CLINICAL TRIAL: NCT04473911
Title: Reduced Intensity Haploidentical Peripheral Blood Stem Cell Transplantation With Post-transplant Cyclophosphamide and Sirolimus/Mycophenolate Mofetil/RGI-2001 Based GVHD Prevention: a Pilot Study
Brief Title: Haplo Peripheral Blood Sct In GVHD Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zachariah Michael DeFilipp (Other)
Collaborators: Regimmune Corporation (Industry)
Responsible Party: Sponsor-Investigator, Zachariah Michael DeFilipp, Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-336
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: GVHD; AML; ALL; MDS; MPN; CMML; Hodgkin Lymphoma; Non Hodgkin Lymphoma; Blood Stem Cell Transplant Failure; Graft Vs Host Disease; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorder; Chronic Myelomonocytic Leukemia; Chemosensitive Hodgkin Lymphoma
Keywords: GVHD; AML; ALL; MDS; MPN; CMML; Hodgkin Lymphoma; Non Hodgkin Lymphoma; Blood Stem Cell Transplant Failure; Graft Vs Host Disease; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorder; Chronic Myelomonocytic Leukemia; Chemosensitive Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Graft vs Host Disease; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Melphalan; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regimen 1: Fludarabine, Cyclophosphamide, and TBI (Experimental): -. Patients who meet eligibility criteria for the study will subsequently be enrolled for treatment. Two reduced intensity regimens will be allowed, according to the choice of the treating physician
  * Pre- stem cell transplant:
    * Fludarabine predetermined dose, intravenously, 4 times per cycle
    * Cyclophosphamide predetermined dose, predetermined number of times in cycle, intravenous infusion
    * Total body irradiation (TBI) once during treatment cycle
  * Post stem cell transplant:
    * Cyclophosphamide predetermined dose, predetermined number of times in cycle, intravenous infusion
    * Sirolimus: Predetermined dosage, predetermined number of time in cycle, oral.
    * Mycophenolate mofetil, oral or iv(predetermined dose or IV TID (based upon actual body weight), at predetermined times per cycle
    * RGI-2001: IV, predetermined dose, weekly to 6 total doses
  Interventions: Drug: FLUDARABINE; Drug: CYCLOPHOSPHAMIDE; Radiation: TBI; Drug: Sirolimus; Drug: Mycophenolate mofetil; Drug: RGI-2001
- Regimen 2: Fludarabine, Melphalan, and TBI (Experimental): -. Patients who meet eligibility criteria for the study will subsequently be enrolled for treatment. Two reduced intensity regimens will be allowed, according to the choice of the treating physician
  * Pre- stem cell transplant:
    * Fludarabine predetermined dose, intravenously 3 times per cycle
    * Melphalan, infusion, determined dosage, once per cycle
    * Total body irradiation (TBI) once per cycle.
  * Post stem cell transplant
    * Cyclophosphamide predetermined dose, predetermined number of times in cycle, intravenous infusion
    * Sirolimus: Predetermined dosage, predetermined number of time in cycle, oral:
    * Mycophenolate mofetil, oral or iv(predetermined dose or IV TID (based upon actual body weight), at predetermined times per cycle
    * RGI-2001: IV, predetermined dose, weekly to 6 total doses
  Interventions: Drug: FLUDARABINE; Radiation: TBI; Drug: Melphalan; Drug: Sirolimus; Drug: Mycophenolate mofetil; Drug: RGI-2001; Drug: CYCLOPHOSPHAMIDE

INTERVENTIONS:
Drug: FLUDARABINE — predetermined dose, intravenously, a predetermined times per cycle Given in both pre stem cell and post stem cell cycles
  Other Names: Fludara®
Drug: CYCLOPHOSPHAMIDE — ◦Cyclophosphamide predetermined dose, predetermined number of times in Given in pre-stem cell Regimen #1 Cyclophosphamide predetermined dose, predetermined number of times in cycle, intravenous infusion
  Other Names: Cytoxan®; Neosar®
  Arms: Regimen 1: Fludarabine, Cyclophosphamide, and TBI
Radiation: TBI — Total body irradiation (TBI) once per cycle.
Drug: Melphalan — Melphalan, infusion, determined dosage, once per cycle
  Other Names: Alkeran®; L-PAM; L-Sarcolysin; Phenylalanine Mustard
  Arms: Regimen 2: Fludarabine, Melphalan, and TBI
Drug: Sirolimus — Sirolimus: Predetermined dosage, predetermined number of time in cycle, oral: Please note that doses of sirolimus can be adjusted at the treating physician's discretion given the multiple drugs and other situations which affect its metabolism
  Other Names: Rapamune
Drug: Mycophenolate mofetil — ◦Mycophenolate mofetil, oral or iv(predetermined dose or IV TID (based upon actual body weight), at predetermined times per cycle
  Other Names: CellCept; Myfortic
Drug: RGI-2001 — IV, predetermined dose, weekly to 6 total doses
Drug: CYCLOPHOSPHAMIDE — ◦Given in Post Stem Cell cycle of Regimen #1 and #2 Cyclophosphamide predetermined dose, predetermined number of times in cycle, intravenous infusion
  Other Names: Cytoxan®; Neosar®

SUMMARY:
This research study is studying the RGI-2001 for preventing Graft-vs-Host Disease (GVHD) in people with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), myelodysplastic syndrome (MDS), myeloproliferative disorders (MPN), chronic myelomonocytic leukemic (CMML), chemosensitive hodgkin lymphoma (HL), or Non-Hodgkin lymphoma (NHL).who will have a blood stem cell transplantation.

* GVHD is a condition in which cells from the donor's tissue attack the organs.
* RGI-2001 is an investigational treatment

DETAILED DESCRIPTION:
* This is a pilot study in subjects undergoing reduced-intensity haploidentical peripheral blood stem cell transplantation who will receive graft-versus-host disease prevention with post-transplant cyclophosphamide, followed by sirolimus, mycophenolate mofetil, and RGI-2001.
* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
* The standard of care drugs of fludarabine, cyclophosphamide, melphalan, radiation, sirolimus, and mycophenolate mofetil are all FDA approved.

  * Eligible Participants will be placed in 1 of 2 groups, per physicians discretion:
  * Regimen #1 :

    * Before stem cell transplant:Fludarabine + Cyclophosphamide + Radiation
    * After stem cell transplant: Cyclophosphamide + Sirolimus +Mycophenolate mofetil + RGI-2001
  * Regimen #2

    * Before stem cell transplant: fludarabine + melphalan + radiation
    * After stem cell transplant: cyclophosphamide + sirolimus +Mycophenolate mofetil + RGI-2001
* A total of 20 participants will be enrolled to this trial
* The U.S. Food and Drug Administration (FDA) has not approved RGI-2001 as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 80 years old
* Diagnosis of hematological malignancy:

  * Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) in morphologic complete remission
  * Myelodysplastic syndrome (MDS), myeloproliferative disorders (MPN), or chronic myelomonocytic leukemic (CMML) with < 5% blasts in blood or bone marrow
  * Chemosensitive Hodgkin lymphoma (HL) or Non-Hodgkin lymphoma (NHL)
* Patients must be undergoing haploidentical allogeneic hematopoietic cell transplantation, defined as 1st or 2nd degree relative with at least 5/10 matching at HLA-A, -B, -C, DR, and DQ.
* ECOG performance status ≤2
* Patients with adequate physical function as measured by:

  * Cardiac: Left ventricular ejection fraction at rest must be ≥ 40%, or shortening fraction >25%
  * Hepatic:

    * Bilirubin ≤ 2.5 mg/dL, except for patients with Gilbert's syndrome or hemolysis
    * ALT, AST, and Alkaline Phosphatase < 5 x ULN
  * Renal: Serum creatinine within normal range, or if serum creatinine is outside normal range, then renal function (measured or estimated creatinine clearance or GFR) ≥ 40mL/min/1.73m2
  * Pulmonary: DLCO (corrected for hemoglobin), FEV1 and FVC ≥ 50% predicted
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplantation. (Patients may have received a prior autologous hematopoietic stem cell transplant.)
* Participants who are receiving any other investigational agents within 14 days prior to RGI-2001 dosing. Thus, participants must stop investigational agents by Day -9 prior to transplant.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, recent myocardial infarction or stroke, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active or uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Planned use of prophylactic donor lymphocyte infusion (DLI) therapy.
* Pregnant and breast-feeding women are ineligible because they are not eligible for hematopoietic stem cell transplantation.
* HIV-positive participants and patients with active Hepatitis B or C are ineligible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving successful donor engraftment | 60 Days
  (absolute neutrophil count > 500/uL and ≥ 90% donor cell chimerism)

SECONDARY OUTCOMES:
100-day non-relapse mortality (NRM) rate. | 100 Days
  The regimen will be considered as safe if 100d NRM rate is <=5%, and not safe if 100d NRM rate is ≥25%.

CONTACTS AND LOCATIONS:
Overall Officials: Zachariah DeFilipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to, please contact the Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation